CLINICAL TRIAL: NCT03647176
Title: PLA Army General Hospital of Beijing
Brief Title: A Comparison of the Resection Rate of Cold Snare Polypectomy for Large (10-15 mm) and Small (5-9 mm) Colorectal Polyps
Acronym: CSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuqi He (Other)
Responsible Party: Sponsor-Investigator, Yuqi He, Principal Investigator, Clinical Professor, General Hospital of Beijing PLA Military Region
Organization: General Hospital of Beijing PLA Military Region (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLA GH-CSP-1
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Adenomatous Polyps
Keywords: Cold snare polypectomy; Colorectal polyps; CARE Study
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- small polyps (Active Comparator): Cold snare polypectomy ; Polyp size will be measured using the tip of the snare catheter (2.5mm).Small (5-9 mm) colorectal polyps will be removed with a polypectomy snare. Following the resection, jet stream of water will be used to wash mucosal defect thoroughly. After endoscopist's attestation that polyp removal was complete by carefully observe the resection margins with near focus mode, biopsies were performed from two marginal sites located symmetrically on the left and right of the mucosal defects to confirm residual polyp tissue.
  Interventions: Other: Cold snare polypectomy
- large polyps (Experimental): Cold snare polypectomy; Polyp size will be measured using the tip of the snare catheter (2.5mm). Large (10-15 mm) colorectal polyps will be removed with a polypectomy snare. Following the resection, jet stream of water will be used to wash mucosal defect thoroughly. After endoscopist's attestation that polyp removal was complete by carefully observe the resection margins with near focus mode, 4 biopsies will be performed from all four quadrants of resection margins.
  Interventions: Other: Cold snare polypectomy

INTERVENTIONS:
Other: Cold snare polypectomy — cold snare polypectomy (CSP), which does not include electrocautery to do a polypectomy with a snare

SUMMARY:
Colorectal cancer remains the third most common cause of death from cancer worldwide. Colonoscopy allows removal of adenomatous polyps is the best colorectal cancer screening, according to the adenoma-carcinoma sequence. Recent studies have reported approximately 30% of interval cancer may be incomplete polyp resection. Complete polyp resection may be particularly important when implementing new methods for surveillance colonoscopies. Cold snare polypectomy (CSP) is considered to be a safer procedure for removing subcentimeter lesions than conventional hot snare polypectomy (HSP). CSP removal of polyps sized ≤5 mm have recommended by the European Society of Gastrointestinal Endoscopy guideline as the preferred technique. Previous report said that the complete resection rate of CSP for adenomatous polyps 4-9 mm in size was comparable to that of HSP, and in the foreseeable future CSP can be one of the standard techniques for 4-9 mm colorectal polyps. However, data on complete resection of colorectal polyps 1.0-1.5 mm in size is sparse. Investigators are interested in comparison of the resection rate of cold snare polypectomy for large (10-15 mm) and small (5-9 mm) colorectal polyps using CSP.

DETAILED DESCRIPTION:
Participantswho meet inclusion criteria will be asked to participate, investigators will include all patients with resectable polyps, but only adenomatous polyps will be included for analysis. See also inclusion and exclusion criteria.

Colonoscopy, after bowel preparation with polyethylene glycol solution was performed using standard colonoscopes (CF-HQ290I, CF-Q260AI) and polypectomy snares(13mm Captivator and 10mm Captivator II).

All procedures were performed by experienced endoscopists (each with over 1000 colonoscopies performed) including CSP. All polyps between 5 and 15mm will be removed with a polypectomy snare. Polyp size will be measured using the tip of the snare catheter (2.5mm). Difficulty of resection will be grade by polyp resection time. Following the resection, jet stream of water will be used to wash mucosal defect thoroughly. After endoscopist's attestation that polyp removal was complete by carefully observe the resection margins with near focus mode, for large lesions (10-15mm) 4 biopsies will be performed from all four quadrants of resection margins, for small lesions (5-9mm) biopsies were performed from two marginal sites located symmetrically on the left and right of the mucosal defects to confirm residual polyp tissue.

If polyp resection is complicated by bleeding (not self-sustained), no biopsies will be taken and any additional polyps that will be found during the remaining examination will be excluded from analysis. Severe bleeding that will complicate resection margins examination will be excluded from analysis, Endoscopic haemostasis will be performed when active haemorrhage continued for ≥30s.

A single research subject may have many eligible polyps. To avoid taking many biopsies, the investigators will not include more than 5 eligible polyps (the first 5 that are detected) per patient in the study.

Laboratory Analysis:

The polyps will be evaluated by experienced pathologists according to Vienna classification. Resection margins for each polyp will be recorded as: R0= adenomatous tissue free, R1=adenomatous tissue detection. Investigators will only include adenomatous polyps in the analysis. for financial requests of the resection margin biopsies. The pathological diagnosis of the biopsies will become part of the medical record. If biopsies contain adenomatous tissue the participants will be ask to return for a follow-up colonoscopy within six month.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥40 and <85
* Provide written informed consent
* Patients are found to have colorectal polyps between 5 and 15mm in size

Exclusion Criteria:

* History of inflammatory bowel disease
* Polyposis of the alimentary tract
* Antiplatelet or anticoagulant therapy 5 days before the procedure
* Pregnancy
* Haemodialysis
* An American Society of Anaesthesiologists class III or higher
* Depressed lesions and lesions highly suspected to be cancerous based on endoscopic appearance

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 40 Years to 85 Years
Enrollment: 1000 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
incomplete CSP resection rate of neoplastic polyps and subgroup analyses of possible factors that could contribute to an incomplete resection | six months
  Incomplete resection was presence of neoplastic tissue from histopathologic examination of polyp margin biopsies. Subgroup included polyp size (5-7mm/8 -9mm/10 -15mm), location (right/left side was defined proximal/distal to the splenic flexure), location with respect to colonic folds (between/on the fold or not), flat morphology (measured by the tip of the 2.4-mm snare catheter), en bloc vs piecemeal resection, a snare exclusively designed as a cold snare versus traditional polypectomy snare, Neoplastic polyps( Adenoma, sessile serrated adenomas/polyps, high-grade dysplasia), and ease of polyp resection (easy or 30s; moderately difficult or 30-60s, difficult or 60s).

SECONDARY OUTCOMES:
polypectomy procedure times | six months
  Time required for resection was defined as the time between the insertion of the snare into working channel to the end of polyp resection
the rates of procedure-related complications | six months
  Delayed bleeding was defined as haemorrhage after colonoscopy requiring endoscopic haemostasis;submucosal disruption; perforation

OTHER OUTCOMES:
adequate assessment of the polyp lateral or vertical margin | 1 year
  Pathological assessment
margins assess after resection | 1 year
  narrow band imaging to delineate polyp margins

CONTACTS AND LOCATIONS:
Overall Officials: tianyang zhang, Principal Investigator — Medical department
Locations (1):
- Department of Gastroenterology, PLA Army General Hospital, Beijing, Dongcheng District, China

IPD SHARING:
Plan to Share IPD: No
individual participant data can be seen after article been published

REFERENCES:
- [Result] Kawamura T, Takeuchi Y, Asai S, Yokota I, Akamine E, Kato M, Akamatsu T, Tada K, Komeda Y, Iwatate M, Kawakami K, Nishikawa M, Watanabe D, Yamauchi A, Fukata N, Shimatani M, Ooi M, Fujita K, Sano Y, Kashida H, Hirose S, Iwagami H, Uedo N, Teramukai S, Tanaka K. A comparison of the resection rate for cold and hot snare polypectomy for 4-9 mm colorectal polyps: a multicentre randomised controlled trial (CRESCENT study). Gut. 2018 Nov;67(11):1950-1957. doi: 10.1136/gutjnl-2017-314215. Epub 2017 Sep 28. PMID 28970290
- [Result] Matsuura N, Takeuchi Y, Yamashina T, Ito T, Aoi K, Nagai K, Kanesaka T, Matsui F, Fujii M, Akasaka T, Hanaoka N, Higashino K, Tomita Y, Ito Y, Ishihara R, Iishi H, Uedo N. Incomplete resection rate of cold snare polypectomy: a prospective single-arm observational study. Endoscopy. 2017 Mar;49(3):251-257. doi: 10.1055/s-0043-100215. Epub 2017 Feb 13. PMID 28192823
- [Derived] Ma X, Feng X, Li Y, Du Y, Wang J, Wu Y, Jin H, Xie X, Wang X, Jin P, Yang L, Wang H, Leung J, Sheng J, He Y. A Comparison of Incomplete Resection Rate of Large and Small Colorectal Polyps by Cold Snare Polypectomy. Clin Gastroenterol Hepatol. 2022 May;20(5):1163-1170. doi: 10.1016/j.cgh.2021.11.010. Epub 2021 Nov 17. PMID 34798334